CLINICAL TRIAL: NCT04879329
Title: A Phase 2 Multi-Cohort, Open-Label, Multi-Center Clinical Study Evaluating the Efficacy and Safety of Disitamab Vedotin (RC48-ADC) Alone or in Combination With Pembrolizumab in Subjects With Locally-Advanced Unresectable or Metastatic Urothelial Carcinoma That Expresses HER2
Brief Title: A Study of Disitamab Vedotin Alone or With Pembrolizumab in Urothelial Cancer That Expresses HER2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC48G001; C5731002 (Other: Alias Study Number); 2022-500030-28-01 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-04-19; First posted 2021-05-10 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial Cancer; Bladder Cancer; HER2 Mutations; HER2 Overexpression; HER2 Amplification; RC48; Seattle Genetics
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — disitamab vedotin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Cohorts A, B, C, D, and G will enroll simultaneously. Cohort E will begin enrollment after Cohort D participants have completed the DLT evaluation period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort A - DV monotherapy for HER2-positive tumor types (Experimental): Disitamab vedotin monotherapy
  Interventions: Drug: disitamab vedotin
- Cohort B - DV monotherapy for HER2-low tumor types (Experimental): Disitamab vedotin monotherapy
  Interventions: Drug: disitamab vedotin
- Cohort C - Non-randomized combination therapy (Experimental): Disitamab vedotin + pembrolizumab
  Interventions: Drug: disitamab vedotin; Drug: pembrolizumab
- Cohort C - Randomized combination therapy (Experimental): Disitamab vedotin + pembrolizumab
  Interventions: Drug: disitamab vedotin; Drug: pembrolizumab
- Cohort C - Randomized monotherapy (Experimental): Disitamab vedotin monotherapy
  Interventions: Drug: disitamab vedotin
- Cohort D - DV monotherapy (Japan only) (Experimental): Disitamab vedotin monotherapy
  Interventions: Drug: disitamab vedotin
- Cohort E - DV combination therapy (Japan only) (Experimental): Disitamab vedotin + pembrolizumab
  Interventions: Drug: disitamab vedotin; Drug: pembrolizumab
- Cohort G - DV monotherapy (Experimental): Disitamab vedotin
  Interventions: Drug: disitamab vedotin

INTERVENTIONS:
Drug: disitamab vedotin — Given into the vein (IV; intravenous) every 2 weeks.
  Other Names: RC48-ADC
Drug: pembrolizumab — Given by IV on Day 1 of each 6-week cycle.
  Other Names: KEYTRUDA®
  Arms: Cohort C - Non-randomized combination therapy; Cohort C - Randomized combination therapy; Cohort E - DV combination therapy (Japan only)

SUMMARY:
This study is being done to see if a drug called disitamab vedotin, alone or with pembrolizumab, works to treat HER2 expressing urothelial cancer. It will also test how safe the drug is for participants.

Participants will have cancer that has spread in the body near where it started (locally advanced) and cannot be removed (unresectable) or has spread through the body (metastatic).

It will also study what side effects happen when participants get the drug. A side effect is anything a drug does to your body besides treating the disease.

ELIGIBILITY:
Inclusion Criteria:

Cohorts A and B

* Histopathologically-confirmed, locally-advanced, unresectable or metastatic urothelial cancer (LA/mUC), including UC originating from the renal pelvis, ureters, bladder, or urethra
* Participants must have received only 1 or 2 lines of prior systemic treatment for LA/mUC, including 1 line of platinum-containing chemotherapy
* At least one measurable lesion by investigator assessment based on RECIST version 1.1.
* HER2-expression status determined by the central laboratory to be IHC 1+, 2+ or 3+, in the provided tumor sample
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Cohort C

* Histopathologically-confirmed LA/mUC, including UC originating from the renal pelvis, ureters, bladder, or urethra
* No prior systemic therapy for LA/mUC

  * Neoadjuvant or adjuvant therapy, including PD-(L)1 inhibitors, is acceptable, if disease recurrence/progression occurred more than 12 months after the last dose of systemic therapy
* At least one measurable lesion by investigator assessment based on RECIST v1.1.
* Participant is eligible to receive cisplatin- or carboplatin- containing chemotherapy per investigator evaluation
* HER2-expression status determined by the central laboratory to be IHC 1+, 2+ or 3+, on the provided tumor tissue sample
* ECOG performance status of 0, 1, or 2

Cohort D

* Histopathologically-confirmed LA/mUC, including UC originating from the renal pelvis, ureters, bladder, or urethra
* Based on a participant's eligibility to receive treatment with standard of care therapies in Japan, participants must have received all of the following lines of therapy for LA/mUC:

  * a. One prior line of platinum-containing chemotherapy.
  * b. Prior therapy with PD-(L)1 inhibitors as (neo)adjuvant therapy, first-line maintenance therapy or as second line treatment.
  * c. Prior enfortumab vedotin therapy.
* At least one measurable lesion by investigator assessment based on RECIST v1.1.
* ECOG performance status of 0 or 1

Cohort E

* Histopathologically-confirmed LA/mUC, including UC originating from the renal pelvis, ureters, bladder, or urethra
* No prior systemic therapy for LA/mUC

  * Neoadjuvant or adjuvant therapy, including PD-(L)1 inhibitors, is acceptable, if disease recurrence/progression occurred more than 12 months after the last dose of systemic therapy.
* At least one measurable lesion by investigator assessment based on RECIST v1.1.
* Participant is eligible to receive cisplatin- or carboplatin- containing chemotherapy per investigator evaluation
* HER2-expression status determined by the central laboratory to be IHC 1+, 2+ or 3+, in the provided tumor sample
* ECOG performance status of 0 or 1

Cohort G

* Histopathologically-confirmed, locally-advanced, unresectable or metastatic urothelial cancer (LA/mUC), including UC originating from the renal pelvis, ureters, bladder, or urethra
* Participants must have received only 1 or 2 lines of prior systemic treatment for LA/mUC, including 1 line of therapy containing enfortumab vedotin as monotherapy or in combination with pembrolizumab

  * The last administration of enfortumab vedotin must be 90 days from the start of study treatment. Intervening therapies are allowed between the final dose of enfortumab vedotin and the start of disitamab vedotin.
* At least one measurable lesion by investigator assessment based on RECIST version 1.1.
* HER2-expression status determined by the central laboratory to be IHC 1+, 2+ or 3+, in the provided tumor sample
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Exclusion Criteria:

Cohorts A and B

* Known hypersensitivity to disitamab vedotin or any of their components
* Prior antitumor treatment (including chemotherapy, radiotherapy, targeted therapy, immunotherapy etc.) within 2 weeks of start of study (defined as Cycle 1 Day 1 for Cohorts A and B)
* Toxicity from a previous treatment has not returned to Grades 0 or 1 (except for Grade 2 alopecia)
* Prior MMAE-based ADCs (eg, enfortumab vedotin) or HER2-directed therapy
* Major surgery that has not fully recovered within 4 weeks prior to dose administration
* Peripheral sensory or motor neuropathy ≥ Grade 2 at baseline

Cohort C

* Known hypersensitivity to disitamab vedotin, pembrolizumab, or any of their components
* Prior antitumor treatment (including chemotherapy, radiotherapy, targeted therapy, immunotherapy etc.) within 2 weeks of start of study defined as Cycle 1 Day 1 for the single-arm part of Cohort C and as randomization date for the randomized part of Cohort C)
* Toxicity from a previous treatment has not returned to Grades 0 or 1 (except for Grade 2 alopecia)
* Prior MMAE-based ADCs (eg, enfortumab vedotin) or HER2-directed therapy
* Major surgery that has not fully recovered within 4 weeks prior to dose administration
* Peripheral sensory or motor neuropathy ≥ Grade 2 at baseline
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug
* Participants who have previously received any prior treatment with an agent directed to another stimulatory or co-inhibitory T cell receptor (including but not limited to CD137 agonists, CAR-T cell therapy, CTLA-4 inhibitors, or OX-40 agonists) are excluded.

Cohort D

* Known hypersensitivity to disitamab vedotin or any of their components
* Prior antitumor treatment (including chemotherapy, radiotherapy, targeted therapy, immunotherapy etc.) within 2 weeks of start of study (defined as Cycle 1 Day 1 for Cohort D)
* Toxicity from a previous treatment has not returned to Grades 0 or 1 (except for Grade 2 alopecia)
* Prior HER2-directed therapy
* Any prior history of ≥ Grade 3 non-hematological AEs related to prior therapy
* Major surgery that has not fully recovered within 4 weeks prior to dose administration
* Peripheral sensory or motor neuropathy ≥ Grade 1 at baseline

Cohort E

* Known hypersensitivity to disitamab vedotin, pembrolizumab, or any of their components
* Prior antitumor treatment (including chemotherapy, radiotherapy, targeted therapy, immunotherapy etc.) within 2 weeks of start of study (defined as Cycle 1 Day 1 for Cohort E)
* Toxicity from a previous treatment has not returned to Grades 0 or 1 (except for Grade 2 alopecia)
* Any prior history of ≥ Grade 3 non-hematological AEs related to prior therapy
* Prior MMAE-based ADCs (eg, enfortumab vedotin) or HER2-directed therapy
* Major surgery that has not fully recovered within 4 weeks prior to dose administration
* Peripheral sensory or motor neuropathy ≥ Grade 1 at baseline
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug

Cohort G

* Known hypersensitivity to disitamab vedotin or any of their components
* Prior antitumor treatment (including chemotherapy, radiotherapy, targeted therapy, immunotherapy etc.) within 2 weeks of start of study (defined as Cycle 1 Day 1 for Cohort G)
* Toxicity from a previous treatment has not returned to Grades 0 or 1 (except for Grade 2 alopecia)
* Prior HER2-directed therapy
* Major surgery that has not fully recovered within 4 weeks prior to dose administration
* Peripheral sensory or motor neuropathy ≥ Grade 2 at baseline

There are additional inclusion and exclusion criteria. The study center will determine if criteria for participation are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2029-04-14 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (cORR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1) by blinded independent central review (BICR) (Cohorts A, B, C, and G) | Duration of treatment; approximately 2 years
  The proportion of participants with confirmed complete response (CR) or partial response (PR) according to RECIST v1.1
Incidence of adverse events (AEs) (Cohorts D and E) | Approximately 2 years
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Incidence of dose alterations (Cohorts D and E) | Approximately 2 years
Incidence of laboratory abnormalities (Cohorts D and E) | Approximately 2 years
  To be summarized using descriptive statistics.
Incidence of electrocardiogram (ECG) abnormalities (Cohorts D and E) | Approximately 2 years
Change from baseline of left ventricular ejection fraction (LVEF) (Cohorts D and E) | Approximately 2 years
Pharmacokinetic (PK) parameter - Area under the curve (AUC) (Cohorts D and E) | Through 30-37 days following the last dose of DV; up to approximately 2 years
  To be summarized using descriptive statistics.
PK parameter - Maximum concentration (Cmax) (Cohorts D and E) | Through 30-37 days following the last dose of DV; up to approximately 2 years
  To be summarized using descriptive statistics.
PK parameter - Time to maximum concentration (Tmax) (Cohorts D and E) | Through 30-37 days following the last dose of DV; up to approximately 2 years
  To be summarized using descriptive statistics.
PK parameter - Trough concentration (Ctrough) (Cohorts D and E) | Through 30-37 days following the last dose of DV; up to approximately 2 years
  To be summarized using descriptive statistics.

SECONDARY OUTCOMES:
cORR per RECIST v1.1 by investigator assessment (Cohorts A, B, C, and G) | Duration of treatment; approximately 2 years
  The proportion of participants with confirmed CR or PR according to RECIST v1.1
Confirmed Duration of Response (DOR) per RECIST v1.1 by BICR (Cohorts A, B, C, and G) | From start of treatment to completion of response assessment; approximately 2 years
  The time from first documentation of objective tumor response (confirmed CR or PR) to the first documentation of tumor progression per RECIST v1.1 or death due to any cause.
Confirmed DOR per RECIST v1.1 by investigator assessment (Cohorts A, B, C, and G) | From start of treatment to completion of response assessment; approximately 2 years
  The time from first documentation of objective tumor response (confirmed CR or PR) to the first documentation of tumor progression per RECIST v1.1 or death due to any cause.
Progression-free survival (PFS) per RECIST v1.1 by BICR (Cohorts A, B, C, and G) | From start of treatment to completion of response assessment; approximately 2 years
  The time from the start of study treatment or randomization (if applicable) to the first documentation of disease progression per RECIST v1.1 or death due to any cause.
PFS per RECIST v1.1 by investigator assessment (Cohorts A, B, C, and G) | From start of treatment to completion of response assessment; approximately 2 years
  The time from the start of study treatment or randomization (if applicable) to the first documentation of disease progression per RECIST v1.1 or death due to any cause.
Disease control rate (DCR) per RECIST v1.1 by BICR (Cohorts A, B, C, and G) | From start of treatment to completion of response assessment; approximately 2 years
  The proportion of participants who have achieved objective response (confirmed CR or PR as per RECIST v1.1 criteria) or stable disease (SD) lasting at least 5 weeks.
DCR per RECIST v1.1 by investigator (Cohorts A, B, C, and G) | From start of treatment to completion of response assessment; approximately 2 years
  The proportion of participants who have achieved objective response (confirmed CR or PR as per RECIST v 1.1 criteria) or SD lasting at least 5 weeks.
Overall survival (OS) (Cohorts A, B, C, and G) | Duration of study; approximately 3 years
  The time from start of study treatment or randomization (if applicable) to the date of death due to any cause.
Incidence of adverse events (AEs) (Cohorts A, B, C, and G) | Approximately 2 years
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Incidence of dose alterations (Cohorts A, B, C, and G) | Approximately 2 years
  To be summarized using descriptive statistics.
Incidence of laboratory abnormalities (Cohorts A, B, C, and G) | Approximately 2 years
  To be summarized using descriptive statistics.
Incidence of ECG abnormalities (Cohorts A, B, C, and G) | Approximately 2 years
Change from baseline of LVEF (Cohorts A, B, C, and G) | Approximately 2 years
PK parameter - AUC (Cohorts A, B, C, and G) | Through 30-37 days following the last dose of DV; up to approximately 2 years
  To be summarized using descriptive statistics.
PK parameter - Cmax (Cohorts A, B, C, and G) | Through 30-37 days following the last dose of DV; up to approximately 2 years
  To be summarized using descriptive statistics.
PK parameter - Tmax (Cohorts A, B, C, and G) | Through 30-37 days following the last dose of DV; up to approximately 2 years
  To be summarized using descriptive statistics.
PK parameter - Ctrough (Cohorts A, B, C, and G) | Through 30-37 days following the last dose of DV; up to approximately 2 years
  To be summarized using descriptive statistics.
PK parameter of pembrolizumab - Cmax (Cohort E) | Through 30-37 days following the last dose of DV; up to approximately 2 years
  To be summarized using descriptive statistics.
Incidence of anti-drug antibodies (ADAs) against disitamab vedotin (All Cohorts) | Through 30-37 days following the last dose of DV; up to approximately 2 years
  To be summarized using descriptive statistics.
Incidence of anti-drug antibodies (ADAs) against pembrolizumab (Cohorts C and E) | Through 30-37 days following the last dose of DV; up to approximately 2 years
  To be summarized using descriptive statistics.
Incidence of neutralizing antibodies (NABs) against disitamab vedotin (All Cohorts) | Through 30-37 days following the last dose of DV; up to approximately 2 years
  To be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (216):
- United States (153):
  - Banner Gateway Medical Center, Gilbert, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Kaiser Permanente Anaheim Kraemer Medical Offices, Anaheim, California
  - Foothill Cardioology, Arcadia, California
  - Kaiser Permanente Baldwin Park Medical Center, Baldwin Park, California
  - Kaiser Permanente Bellflower Medical Offices, Bellflower, California
  - Beverly Hills Multi-Specialties Practice, Beverly Hills, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - UCLA Burbank Cardiology, Burbank, California
  - UCLA Hematology/Oncology - Burbank, Burbank, California
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - UCLA Encino Specialty Care (Radiology), Encino, California
  - UCLA Hematology/Oncoclogy-Encino, Encino, California
  - Kaiser Permanente Fontana Medical Center, Fontana, California
  - Foothill Cardiology Glendora, Glendora, California
  - Kaiser Permanente South Bay Medical center, Harbor City, California
  - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Kaiser Permanente Alton/Sand Canyon Medical Offices, Irvine, California
  - UCLA Downtown Los Angeles Primary & Specialty Care, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Offices, Los Angeles, California
  - Kaiser Permanente West Los Angeles Medical Center, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - UCLA Cardiovascular Center, Los Angeles, California
  - UCLA Hematology Oncology, Los Angeles, California
  - UCLA Westwood Specialty Care, Los Angeles, California
  - UCLA Santa Monica Cardiology, Los Angeles, California
  - UCLA Montecito Primary & Specialty Care, Montecito, California
  - Newport Diagnostics Center (Radiology), Newport Beach, California
  - Kaiser Permanente Ontario Medical Center, Ontario, California
  - UC Irvine Health, Orange, California
  - Kaiser Permanente Panorama City Medical Center, Medical Offices 3, Panorama City, California
  - Foothill Cardiology Pasadena, Pasadena, California
  - Southern California Heart Specialists, Pasadena, California
  - UCLA Hematology/ Oncology- Pasadena, Pasadena, California
  - UCLA Hematology Oncology - Porter Ranch, Porter Ranch, California
  - UCLA Porter Ranch Primary & Specialty Care, Porter Ranch, California
  - Kaiser Permanente Riverside Medical Center, Riverside, California
  - Southern California Permanente Medical Group (SCPMG), Riverside, California
  - Kaiser Permanente San Diego Mission Road (Regulatory and Lab Supplies), San Diego, California
  - Kaiser Permanente Zion Medical Center, San Diego, California
  - UCSF Cancer Center MZ Phlebotomy, San Francisco, California
  - UCSF Mount Zion Phlebotomy, San Francisco, California
  - UCSF Parnassus Phlebotomy, San Francisco, California
  - UCSF Investigational Drugs Pharmacy, San Francisco, California
  - University of California, San Francisco | HDFCCC - Hematopoietic Malignancies, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Diagnostic Medical Group of Southern California (Radiology), San Gabriel, California
  - Southern California Heart Centers, San Gabriel, California
  - UCLA Hematology/Oncology - San Luis Obispo, San Luis Obispo, California
  - Sierra Vista Regional Medical Center, San Luis Obispo, California
  - Kaiser Permanente San Marcos Medical Offices, San Marcos, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - UCLA Simi Valley Alamo Specialty Care, Simi Valley, California
  - Twin Cities Community Hospital, Templeton, California
  - UCLA Thousand Oaks Primary & Specialty Care, Thousand Oaks, California
  - UCLA Hematology/Oncology - Torrance, Torrance, California
  - UCLA Torrance Lomita Specialty Care, Torrance, California
  - UCLA Hematology-Oncology Clinic - Santa Clarita, Valencia, California
  - UCLA Santa Clarita Primary & Specialty Care, Valencia, California
  - UCLA Hematology/Oncology - Ventura, Ventura, California
  - UCLA Ventura Cardiology, Ventura, California
  - UCLA Hematology/Oncology - Westlake, Westlake Village, California
  - Kaiser Permanente Woodland Hills Medical Center, Woodland Hills, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Bonita Springs, Florida
  - Florida Cancer Specialists, Bradenton, Florida
  - Florida Cancer Specialists, Cape Coral, Florida
  - Florida Cancer Specialists, Daytona Beach, Florida
  - Florida Cancer Specialists, Fleming Island, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, N. Venice, Florida
  - Florida Cancer Specialists, Naples, Florida
  - Florida Cancer Specialists, Port Charlotte, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists, Stuart, Florida
  - Florida Cancer Specialists, Tallahassee, Florida
  - Moffitt Cancer Center McKinley Hospital, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists, Venice, Florida
  - Florida Cancer Specialists, Vero Beach, Florida
  - Florida Cancer Specialists, Wellington, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Northwest Georgia Oncology Centers, a Service of Tanner Medical Center Villa Rica, Carrollton, Georgia
  - West Georgia Infusion Center, a Service of Tanner Medical Center Villa Rica, Carrollton, Georgia
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Cartersville, Georgia
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Douglasville, Georgia
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Hiram, Georgia
  - WellStar Paulding Hospital, Hiram, Georgia
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Marietta, Georgia
  - UChicago Medicine - River East, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Accellacare - Deerfield, Deerfield, Illinois
  - UChicago Medicine at Ingalls - Flossmoor, Flossmoor, Illinois
  - UChicago Medicine Ingalls Memorial, Harvey, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - The University of Chicago Medicine Center for Advanced Care Orland Park, Orland Park, Illinois
  - UChicago Medicine at Ingalls - Tinley Park, Tinley Park, Illinois
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - The Cancer & Hematology Centers, Big Rapids, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Cancer - Detroit (Brigitte Harris Cancer Pavilion), Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - The Cancer & Hematology Centers, Grand Rapids, Michigan
  - Cancer & Hematology Centers of Western Michigan, PC- Kit Storage, Grand Rapids, Michigan
  - The Cancer & Hematology Centers, Holland, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - The Cancer & Hematology Centers, Norton Shores, Michigan
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - MSK Bergen, Montvale, New Jersey
  - MSK Commack, Commack, New York
  - MSK Wesrchester, Harrison, New York
  - Northwell Health, Lake Success, New York
  - Memorial Sloan Kattering Cancer Centre- Investigational Drug Service Pharmacy, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care (74th Street)., New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Evelyn H. Lauder Breast and Imaging Centre (BAIC), New York, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - Sidney Kimmel Center for Prostate and Urological Cancers - Memorial Sloan Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - MSK nassau, Uniondale, New York
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - UNC Lineberger Comprehensive Cancer Center / University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center (biopsy only), Charlotte, North Carolina
  - Carolinas Medical Center Investigational Drug Services, Charlotte, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Mercy (biopsy only), Charlotte, North Carolina
  - Atrium Health University City (biopsy only), Charlotte, North Carolina
  - Levine Cancer Institute University, Charlotte, North Carolina
  - Levine Cancer Institute - Ballantyne, Charlotte, North Carolina
  - Atrium Health Cabarrus (biopsy only), Concord, North Carolina
  - Levine Cancer Institute Concord, Concord, North Carolina
  - Levine Cancer Institute- Gaston, Gastonia, North Carolina
  - Atrium Health Union (biopsy only), Monroe, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - James Cancer Hospital & Solove Research Institute, Columbus, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - OSU Wexner Medical Center & James Cancer Hospital, Columbus, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - OU Medical Center, Oklahoma City, Oklahoma
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baylor Scott and White Research Institute, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - Huntsman Cancer Institute at The University of Utah, Salt Lake City, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Froedtert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (8):
  - Centro de Investigaciones Médicas y Desarrollo LC S.R.L, Buenos Aires, Buenos Aires F.D.
  - Clinica Viedma, Viedma, Río Negro Province
  - Hospital Aleman, Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Buenos Aires
  - Hospital Sirio Libanes - Buenos Aires, Buenos Aires
  - Centro Medico Austral, CABA
  - Centro Oncologico Korben, Caba
  - Instituto Oncologico de Cordoba, Córdoba
- Australia (7):
  - Cancer Care Research Pty Ltd (trading as GenesisCare), Alexandria, New South Wales
  - GenesisCare - North Shore, St Leonards, New South Wales
  - Macquarie University, Sydney, New South Wales
  - Metro South Hospital and Health Service, Brisbane, Queensland
  - Mater Cancer Care Centre, Mater Misericordiae Limited, South Brisbane, Queensland
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Lyell McEwin Hospital, Elizabeth Vale
- Belgium (2):
  - AZ Maria Middelares, Ghent
  - CHU UCL Namur-Site de Saint Elisabeth, Namur
- Canada (6):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - BC Cancer - Vancouver Fairmont Medical Building, Vancouver, British Columbia
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Jewish General Hospital, Montreal, Quebec
  - Centre integre universitaire de sante et de services sociaux de l'Estrie, Sherbrooke, Quebec
- Chile (3):
  - Centro de Estudios Clínicos IC La Serena Research, La Serena, Coquimbo Region
  - Oncovida SA, Santiago, Providencia
  - Pontificia Universidad Catolica de Chile, Santiago, Providencia
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Rabin medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Ospedale San Raffaele, Milan, Lombardy
  - Centro di Riferimento Oncologico Di Aviano, Aviano, Pordenone
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, ROME
  - IRCCS Ospedale San Raffaele, U.O. Farmacia Studi Clinici, Milan
  - IOV-Istituto Oncologico Veneto IRCCS-U.O. Oncologia Medica 1-SC Farmacia, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Ospedaliera S. Maria di Terni, Terni
  - S.C. Farmacia Interna, Terni
- Japan (6):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Osaka University Hospital, Suita-shi, Osaka
  - Tokushima University Hospital, Tokushima, Tokushima
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Osaka Prefectural Hospital Organization - Osaka International Cancer Institute, Osaka
- Spain (5):
  - Hospital Universitari Parc Tauli Sabadell, Sabadell, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - MD Anderson Cancer Center - Madrid, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Turkey (Türkiye) (4):
  - Ankara Universitesi Tip Fakultesi Hastaneleri - Cebeci Arastirma ve Uygulama Hastanesi, Ankara
  - Trakya Universitesi Tip Fakultesi Hastanesi (Saglik Arastirma ve Uygulama Merkezi), Edirne
  - T.C. Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Izmir Ekonomi Universitesi Medical Point Hastanesi, Izmir
- United Kingdom (8):
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Barts Health NHS Trust, St Bartholomew's Hospital, London
  - Guy's Hospital, London
  - Charing Cross Hospital, London
  - The Christie NHS Foundation Trust - Christie Hospital, Manchester
  - The Christie NHS Foundation Trust, Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, The Clatterbridge Cancer Centre - Wirral, Merseyside

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=RC48G001